CLINICAL TRIAL: NCT04679389
Title: A Randomized, Double-blind, Placebo-controlled Study Evaluating Acetazolamide Efficacy in Ataxia in PMM2-CDG
Brief Title: Acetazolamide Efficacy in Ataxia in PMM2-CDG
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Mayo Clinic (Other)
Collaborators: Seattle Children's Hospital (Other); Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Eva Morava-Kozicz, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-000634
Record Dates: First submitted 2020-12-14; First posted 2020-12-22 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Pmm2-CDG; CDG1A
MeSH Terms: conditions — Congenital disorder of glycosylation type 1A | interventions — Gelatin; Lactose; Acetazolamide

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, placebo controlled, with optional extension period
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetazolamide (Experimental): Acetazolamide administered via capsule or liquid suspension. Capsule would be 250 mg oral capsules encapsulated by gelatin capsule and filled with lactose to match placebo. Liquid suspension would be 25 mg/mL oral suspension but adding 125 mg Acetazolamide tablets to suspending agent Ora-blend
  Interventions: Drug: Acetazolamide
- Placebo (Placebo Comparator): Placebo administered via capsule or liquid suspension. Capsule would be a gelatin capsule filled with lactose powder to match Acetazolamide. Liquid suspension would be Ora-blend.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — administered orally or enterally
  Other Names: Gelatin, lactose, and Ora-blend
  Arms: Placebo
Drug: Acetazolamide — administered orally or enterally
  Other Names: Diamox
  Arms: Acetazolamide

SUMMARY:
Objective 1 (Primary): To determine the efficacy of acetazolamide in improving ataxia in patients with PMM2-CDG.

Objective 2 (Secondary): To evaluate for any adverse events related to longer term acetazolamide administration.

Objective 3 (Secondary): To examine the effect of acetazolamide on PMM2 biomarkers including carbohydrate deficient transferrin results, electrolytes (Na, K, Cl, CO2), VBG (pH, pCO2, PO2, CO2, Base excess), liver function tests (AST, ALT, GGT, indirect and direct bilirubin, total protein, albumin, alkaline phosphatase), kidney function tests (BUN, Creatinine, Urinalysis, urine calcium/creatinine ratio, urine protein/creatinine ratio), growth (height, weight, head circumference), vital signs (blood pressure, respiratory rate, heart rate), PROMIS scores, dysarthria using the PATA score, and NPCRS score.

Objective 4 (Secondary): To explore characteristics of individuals with PMM2-CDG who do not respond to acetazolamide.

DETAILED DESCRIPTION:
This study is double-blind, placebo-controlled, 1:1 randomized clinical therapeutic trial of acetazolamide for the treatment of ataxia in patients with PMM2-CDG. Clinical history and screening data will be reviewed to determine subject eligibility. Potential subjects who have a molecularly and/or biochemical confirmed diagnosis of PMM2-CDG will be consented. Baseline data will be collected prior to randomization and at treatment initiation. Subjects who meet all inclusion criteria and none of the exclusion criteria will be enrolled into the study. Each subject who meets all the inclusion and none of the exclusion criteria will then be randomized to placebo or acetazolamide. They will be administered weight-dependent doses of acetazolamide or an equivalent volume of placebo twice daily by mouth. Initial dose of acetazolamide is 8 mg/kg/day if subjects are taking the liquid formulation, or as per Table 1b if they are taking the capsule formulation. If taking the liquid formulation, the dose of study drug will be increased by 7 mg/kg/day to a maximum of 22 mg/kg/day (not to exceed 1000 mg/day) if well tolerated with no treatment related SAEs or abnormal pH. If the pH is <7.32, the dose will be reduced by 7 mg/kg/day. The dose will be adjusted similarly according to Table 1b if taking the capsule formulation. Subjects will be randomized after Visit 1, will initiate blinded therapy within the first week, and will continue on prescribed/adjusted blinded treatment until Visit 4. Of note, the concentration of the liquid formulation and the amount of milligrams of acetazolamide per capsule will stay constant, and the volume or number of capsules will be adjusted based on tolerance as assessed by symptoms and laboratories. If an individual is randomized to the placebo arm, the initial volume will be equivalent to 7 mg/kg/day or the initial number of capsules as per Table 1, and volume or number of capsules will also be adjusted based on symptoms and laboratory values each time dose adjustment is planned. Open label period will then begin after Visit 4 up to Visit 9 (see Figure 1 and Table 3). As both the subject and investigator do not know if the subject received placebo or acetazolamide, the dose of acetazolamide will be started at Visit 4 at 8 mg/kg/day and titrated upwards in the same manner in Visits 5 and 6 (remote) as in Visits 2 and 3 (remote). Subjects will have the option to withdraw from the study any time after Visit 4 if they do not wish to proceed onto or continue with the open label phase.

ELIGIBILITY:
Inclusion Criteria:

* Molecularly and/or enzymatically-confirmed PMM2-CDG,
* Age ≥4 years old, and
* Affected with ataxia evidenced by mini International Cooperative Ataxia Rating Scale (Mini-ICARS) score >0 at baseline.

Exclusion Criteria:

* Hepatic impairment defined as AST/ALT >5x ULN in the last 12 months
* Renal impairment defined as serum creatinine: > 0.5 mg/dL (<6 years); > 0.7 mg/dL (7-10 years); > 1.24 mg/dL (> 11 years)- Hypersensitivity to acetazolamide
* Hypersensitivity to any of the components of the placebo
* History of treatment with experimental drug within 28 days of Visit 1
* Currently taking Mecamylamine, Sodium Phosphates, Salicylates, Mefloquine, Methenamine and other Carbonic Anhydrase Inhibitors

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Morava-Kozicz, MD, PhD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
De-identified data may be shared amongst member of the consortium FCDGC and with the NIH.

RESULTS

PARTICIPANT FLOW:
Groups:
- Acetazolamide: Acetazolamide was administered via capsule or liquid suspension. Capsule was 250 mg oral capsules encapsulated by gelatin capsule and filled with lactose to match placebo. Liquid suspension was 25 mg/mL oral suspension but adding 125 mg Acetazolamide tablets to suspending agent Ora-blend
  Acetazolamide: administered orally or enterally
- Placebo: Placebo was administered via capsule or liquid suspension. Capsule was a gelatin capsule filled with lactose powder to match Acetazolamide. Liquid suspension was a Ora-blend.
  Placebo: administered orally or enterally
Period: Overall Study
Arm/Group | Acetazolamide | Placebo
Started | 13 | 12
Completed | 2 | 0
Not Completed | 11 | 12
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Physician Decision | 3 | 5
Not completed — Withdrawal by Subject | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetazolamide | Placebo | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.62 (8.47) | 10.88 (5.26) | 12.30 (7.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 8 | 10 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 11 | 21
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Acetazolamide on Ataxia Measured Via Miniature International Cooperative Ataxia Rating Scale (Mini-ICARS)
Description: To achieve this goal, we compared the change of Mini-ICARS score from baseline to after six months of treatment between the placebo and active treatment groups. Minimal score is 0, maximum score is 100, higher score indicates greater impairment. Each subscale has an ordinal scale with a 0 indicating normal and the higher score indicating greater impairment or that the patient was unable to complete the task.
Time Frame: baseline-6 months
Population: Data was not collected nor analyzed for two subjects in the Acetazolamide arm and one subject in the Placebo arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 11 | 11
score on a scale | 1.64 (3.20) | 1.36 (3.23)
Statistical Analysis 1: Comparison: Acetazolamide vs Placebo; Test type: Superiority; p = 0.84, t-test, 2 sided

2. Secondary Outcome: Abnormal Blood pH Value
Description: Blood pH level was assessed through venous blood gas test. The number of participants who experience a drug related adverse event related to abnormal blood pH value.
Time Frame: through study completion, approximately 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 13 | 12
Participants | 0 | 1
Statistical Analysis 1: Comparison: Acetazolamide vs Placebo; Test type: Superiority; p = 0.48, Fisher Exact

3. Secondary Outcome: Electrolyte Balance Testing
Description: Electrolyte balance was assessed through combination testing on concentration of potassium, sodium, chloride, bicarbonate, magnesium, calcium, and phosphate. The number of participants who experience a drug related adverse event related to abnormal electrolyte balance.
Time Frame: through study completion, approximately 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 13 | 12
Participants | 0 | 1
Statistical Analysis 1: Comparison: Acetazolamide vs Placebo; Test type: Superiority; p = 0.48, Fisher Exact

4. Secondary Outcome: Urine Calcium Excretion Testing
Description: Urine calcium excretion is measured by mg excreted per day. The number of participants who experience a drug related adverse event related to abnormal excretion of calcium.
Time Frame: through study completion, approximately 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 13 | 12
Participants | 0 | 0
Statistical Analysis 1: Comparison: Acetazolamide vs Placebo; Test type: Superiority; p > 0.99, Fisher Exact

5. Secondary Outcome: Examine Effect of Acetazolamide on PMM2 Biomarker Carbohydrate Deficient Transferrin
Description: Number of patients with abnormal ratio result will be recorded to understand the effect acetazolamide has on this biomarker
Time Frame: 6 months
Population: Data was not collected nor analyzed for this outcome measure. Data collection for this outcome never occurred. PMM2 biomarker carbohydrate deficient transferrin was not collected for any subjects. The test was never collected for any subjects.
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS) Score
Description: PROMIS = Physical activity 10-items from 1(no days) to 5(6-7 days), Strength impact 12-item from 1(no days) to 5(6-7 days), Fatigue 23-item from 1(never) to 5(almost always), Mobility 23-item from 1(not able to do) to 5(with no trouble), Pain interference 13-item from 1(never) to 5(almost always), Upper extremity coordination 29-item from 1(not able to do) to 5(with no trouble), Global Health 9-item from 1(poor) to 5( excellent), Parent Proxy Mobility 8-item from 1(not able to do) to 5(with no trouble), Anxiety 8-item from 1(never) to 5(almost always), Depresson 8-item from 1(never) to 5(almost always), Parent Proxy Fatigue 8-item from 1(never) to 5(almost always), Peer relationships 8-item from 1(never) to 5(almost always), Parent proxy pain interference 8-item from 1(never) to 5(almost always), Pain intensity 1-item from 0(no pain) to 10(worst pain). Total scores range from 168 - 845. Lower scores indicate worse health, higher scores indicate better health
Time Frame: baseline, 6 months
Population: Data was not collected nor analyzed for seven subjects in the Acetazolamide arm and four subjects in the Placebo arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 6 | 8
score on a scale | 3.02 (4.45) | 0.75 (4.09)

7. Secondary Outcome: Change in Dysarthria as Measured by the PATA Score
Description: PATA test measures the number of times a patient can say the word "PATA" in a 10 second time period. Number of "PATA"s spoken in 10 seconds indicates level of dysarthria. The higher the score the less dysarthria, the lower the score more dysarthria.
Time Frame: baseline, 6 months
Population: Data was not collected nor analyzed for four participants in the Acetazolamide arm and three participants in the Placebo arm
Measure: Mean (Standard Deviation); unit: words/10 sec
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 9 | 9
words/10 sec | 2.30 (3.71) | 0.59 (3.11)
Statistical Analysis 1: Comparison: Acetazolamide vs Placebo; Test type: Superiority; p = 0.31, t-test, 2 sided

8. Secondary Outcome: Change in Nijmegen Pediatric CDG Rating Scale (NPCRS)
Description: The NPCRS is a scale that evaluates the patient's current function, system specific involvement, and current clinical assessment. Total scores range from 0 - 82. A mild score is 0-14, moderate score is 15-25, and severe is a score >26.
Time Frame: baseline, 6 months
Population: Data was not collected nor analyzed for three participants in the Acetazolamide arm and one participant in the Placebo arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 10 | 11
score on a scale | 1.20 (1.99) | 0.27 (1.79)
Statistical Analysis 1: Comparison: Acetazolamide vs Placebo; Test type: Superiority; p = 0.09, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 3 years
Arm/Group | Acetazolamide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/13 | 3/12
Other Adverse Events (participants affected / at risk) | 9/13 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetazolamide (N=13) | Placebo (N=12)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Thromboembolic Event (Vascular disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetazolamide (N=13) | Placebo (N=12)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood and Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Ear and Labyrinth Disorders - Other (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eye Disorders - Other (Eye disorders) | 1 (1) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Fatigue (General disorders) | 1 (1) | 3 (5)
Fever (General disorders) | 2 (2) | 2 (3)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 4 (8) | 2 (5)
General Disorders and Administration Site Conditions - Other (General disorders) | 2 (12) | 3 (6)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Immune System Disorders - Other (Immune system disorders) | 1 (1) | 0 (0)
Infections and Infestations - Other (Infections and infestations) | 1 (1) | 5 (6)
Investigations - Other (Investigations) | 0 (0) | 1 (4)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Metabolism and Nutrition Disorders - Other (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Musculoskeletal and Connective Tissue Disorder - Other (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (General disorders) | 1 (1) | 1 (1)
Nervous System Disorders - Other (Nervous system disorders) | 1 (1) | 2 (5)
Otitis Media (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Renal and Urinary Disorders - Other (Renal and urinary disorders) | 3 (3) | 1 (2)
Respiratory, Thoracic and Mediastinal Disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin and Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary Frequency (Renal and urinary disorders) | 4 (4) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 4 (6)
Edema Limbs (General disorders) | 0 (0) | 1 (1)
Rhinitis Infective (Infections and infestations) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT04679389/Prot_SAP_000.pdf